CLINICAL TRIAL: NCT03857412
Title: Evaluation of Intraoperative Capsular Polishing on Lens Epithelial Cells and the Development of Posterior Capsule Opacification
Brief Title: Posterior Capsule Opacification After Lens Capsule Polishing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principle Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Polishing
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Posterior Capsule Opacification
Keywords: Polishing; Cataract surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non capsular polishing (Sham Comparator): No capsular polishing taking place during cataract surgery
  Interventions: Other: Non capsular polishing
- Capsular polishing (Active Comparator): Capsular polishing taking place during cataract surgery
  Interventions: Procedure: Capsular polishing

INTERVENTIONS:
Procedure: Capsular polishing — Capsular polishing taking place during cataract surgery
  Arms: Capsular polishing
Other: Non capsular polishing — No capsular polishing taking place during cataract surgery
  Arms: Non capsular polishing

SUMMARY:
Investigate the effect of polishing of the lens capsule during cataract surgery on the development of posterior capsule opacification

DETAILED DESCRIPTION:
Cataract, the clouding if the eye's lens, is the leading cause of blindness worldwide, with phacoemulsification and implantation of an intraocular lens being the only therapeutic option. Cataract surgery is nowadays considered a safe and efficient procedure. However, one of the most frequent complications after surgery is posterior capsule opacification (PCO), that results in diminished postoperative visual acuity. PCO occurs due to remaining lens epithelial cells in the capsular bag, that start to migrate and proliferate.

PCO can be easily treated by performing a neodymium-doped yttrium aluminium garnet (Nd-YAG) laser capsulotomy. However, even if laser capsulotomy is considered a simple procedure, possible complications are rise of intraocular pressure, inflammation, cystoid macular edema, or retinal detachment. Furthermore, several patients are no suitable candidates for laser capsulotomy, for example children and patients with high myopia.

Therefore, it would be necessery to identify different approaches to prevent generation of PCO. One approach could be "cleaning" of the lens epithelial cells in the capsular bag by polishing of the lens capsule during surgery. Hence, the aim of this study is to examine whether capsular polishing is beneficial to decrease the growth and proliferation of LECs.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract.
* Patients in the age group of 21 years and above.
* Patients with uncomplicated cataract.
* Patients without any relevant systemic or ocular morbidity.
* Patients with well dilating pupils.
* Written informed consent prior to any study specific action.

Exclusion Criteria:

* Patients with complicated cataract.
* Patients having corneal pathology.
* Patients with any form of ocular inflammation.
* Patients with glaucoma, retinal pathologies.
* Patients with traumatic cataracts, subluxated and dislocated lens, prior h/o ocular surgery, pseudoexfoliation.
* Any intraoperative complications like posterior capsule rupture.
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between eye with capsular polishing and eye without capsular polishing concerning generation of posterior capsule opacification (PCO) in the same patient | 6 months
  Posterior capsule opacification will be graded using a score from 0 (clear capsule) to 10 (very severe PCO)

SECONDARY OUTCOMES:
Difference in the number of cells in the anterior chamber between the eye with capsular polishing and the eye without capsular polishing in the same patient | 6 months
  Number of cells in the anterior chamber will be rated using a laser flare meter

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided